CLINICAL TRIAL: NCT00148668
Title: A Randomized Phase II Study of Preoperative Herceptin/Navelbine Versus Taxotere/Carboplatin/Herceptin in Early Stage, HER-2 Positive Breast Cancer
Brief Title: Preoperative Herceptin/Navelbine Versus Taxotere/Carboplatin/Herceptin in HER-2 Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eric Winer, MD (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Yale University (Other)
Responsible Party: Sponsor-Investigator, Eric Winer, MD, Chief Division of Women's Cancers, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-311
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer
Keywords: HER-2 Positive Breast Cancer; herceptin; navelbine; taxotere; carboplatin; Early stage Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Vinorelbine; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Herceptin/navelbine
  Interventions: Drug: Herceptin; Drug: Navelbine
- Arm 2 (Active Comparator): Taxotere/carboplatin/herceptin
  Interventions: Drug: Herceptin; Drug: Taxotere; Drug: Carboplatin

INTERVENTIONS:
Drug: Herceptin — One dose given followed by an MRI, then weekly injections beginning week 3 and ending week 14.
  Other Names: Trastuzumab
Drug: Navelbine — Weekly injections given starting week 3 and ending week 14
  Other Names: vinorelbine
  Arms: Arm 1
Drug: Taxotere — Given every three weeks starting week 3 and ending on week 14
  Other Names: docetaxel
  Arms: Arm 2
Drug: Carboplatin — Given every three weeks starting week 3 and ending on week 14
  Other Names: paraplatin
  Arms: Arm 2

SUMMARY:
The purpose of this study is to find out what effects the preoperative combination therapies of herceptin/navelbine or herceptin/taxotere/carboplatin will have on patients with early stage HER-2 positive breast cancer.

DETAILED DESCRIPTION:
Before starting treatment, a clip will be placed via catheter into the tumor bed, so the surgeon can locate the site of the tumor. During clip placement, tissue biopsy will be taken of the tumor. One to two weeks after the first dose of herceptin another biopsy will be performed.

Patients will be placed into one of 2 arms.

* Arm 1 receives 12 weeks of herceptin and navelbine. Arm 2 receives 4 cycles of taxotere/carboplatin/herceptin.
* Arm 2 participants will also receive neulasta (growth factor support) on day 2 of each cycle.

Phase A of Arm 1 is one dose of herceptin followed by an MRI of the affected breast and a second biopsy 1-2 weeks following this dose. Phase B of Arm 1 begins on week 3 and ends on week 14 and involves weekly injections of herceptin and navelbine. Surgery will take place a minimum of 3 weeks after the patients last dose of herceptin and navelbine.

Phase A of Arm 2 is one dose of herceptin followed by an MRI of the affected breast and second biopsy 1-2 weeks following this dose. Phase B of Arm 2 begins on week 3 and ends on week 14 and involves herceptin weekly, taxotere and carboplatin every 3 weeks. Surgery will take place a minimum of 3 weeks after the patients last dose of herceptin, taxotere and carboplatin.

Blood tests will be performed every 3 weeks during pre-operative treatment and every 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage II or III breast cancer
* HER-2 positive tumors
* Older than 18 years of age
* Eastern Cooperative Oncology Group (ECOG) Performance Status of greater or equal to 1.
* ANC > 1,500/mm3
* Hemoglobin > 9gm/dl
* Platelets > 100,000mm3
* Creatinine < 2mg/dl
* Glucose < 200mg/dl
* Bilirubin < 1.5 x ULN

Exclusion Criteria:

* Previous treatment with herceptin, taxanes, doxorubicin or other anthracycline-type therapy, navelbine, or platinum-based therapy.
* Pregnant or breast-feeding women
* Serious illness, or medical or psychiatric condition
* Uncontrolled infections
* Active or severe cardiovascular or pulmonary disease
* Patients with left ventricular ejection fraction < 50%
* Peripheral neuropathy of any etiology that exceeds grade 1
* Prior history of malignancy
* Uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2003-12; Primary Completion 2009-01 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Winer, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Yale Cancer Center, New Haven, Connecticut
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 81 patients were enrolled on the study between 12/2003 and 8/2008.
Groups:
- Herceptin/Navelbine: Herceptin( 2mg/kg)navelbine (25mg/kg2) x 12 weeks
- Taxotere/Carboplatin/Herceptin: Taxotere (75mg/kg2)/carboplatin (AUC6)/herceptin(2mg/kg)[TC q 3 weeks/H q 1 wk) x 4 cycles
Period: Overall Study
Arm/Group | Herceptin/Navelbine | Taxotere/Carboplatin/Herceptin
Started | 41 | 40
Completed | 41 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 41 | 40 | 81
Age Continuous [Mean (Standard Deviation); unit: years] | 47.8 (12.6) | 48.1 (8.5) | 48 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 40 | 81
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 40 | 81

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response After Preoperative Therapy With Herceptin/Navelbine Versus Taxotere/Carboplatin/Herceptin in Patients With HER-2 Positive Early Breast Cancer
Description: Pathological Complete Response is defined as the complete disappearance of invasive tumor in the breast at the time of surgery
Time Frame: 12 weeks
Population: Please Note that in Arm 2, the number of participants analyzed is equal to 39, which differs from the Number of Participants reported in the baseline measure (N= 40) because one participant withdrew her consent, so was not evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 41 | 39
percentage of participants | 17 | 31

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 5/41 | 5/40
Other Adverse Events (participants affected / at risk) | 27/41 | 25/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=41) | Arm 2 (N=40)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
SGPT (ALT) (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=41) | Arm 2 (N=40)
Leukocytes (Immune system disorders) | 6 (6) | 7 (7)
Neutropenia (Immune system disorders) | 11 (11) | 5 (5)
Febrile Neutropenia (Immune system disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
SGOT (AST) (Hepatobiliary disorders) | 3 (3) | 0 (0)
SGPT (ALT) (Hepatobiliary disorders) | 4 (4) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dehydration (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Irregular Menses (Reproductive system and breast disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No